CLINICAL TRIAL: NCT04841629
Title: Perception & Acceptability of a Cervical Cancer Prevention Prebiotic Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glyciome, LLC (Industry)
Collaborators: Brigham and Women's Hospital (Other); University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: R41CA254543 (NIH)
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Sensory Perceptual Characteristics; User Acceptability of Gel Delivery System

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PreBioGyn Gel (Experimental): Topical administration to forearm
  Interventions: Other: PreBioGyn Gel
- Trimosan Gel (Active Comparator): Topical administration to forearm
  Interventions: Other: Trimosan Gel
- RepHresh Gel (Active Comparator): Topical administration to forearm
  Interventions: Other: RepHresh Gel

INTERVENTIONS:
Other: PreBioGyn Gel — Cellulose-based prebiotic gel developed to optimize vaginal health and reduce the risk of cervical cancer in women.
  Arms: PreBioGyn Gel
Other: Trimosan Gel — Carbomer-based gel
  Arms: Trimosan Gel
Other: RepHresh Gel — Carbomer-based gel
  Arms: RepHresh Gel

SUMMARY:
PreBioGyn will be compared to market leading vaginal pH buffering gels using established forearm test methods associated with vaginal lubricity sensation in 42 women. Women will also rate each gel for smell and appearance using established methods. The PreBioGyn gel enclosure and intravaginal applicator design will be evaluated for: look and feel, ability to prepare for dosing, ability to expulse dose, and likelihood of future use by subjects. Open-ended feedback on the gel and applicator will occur to gather contributions for each product.

DETAILED DESCRIPTION:
This study is being conducted as a component of a NIH/NCI sponsored Small Business Technology Transfer (STTR) project entitled "Cervical Cancer Prevention Prebiotic Device."

The prebiotic vaginal gel, PreBioGyn, has been developed to optimize vaginal health and reduce the risk of cervical cancer in women. Use of the gel targets a combination of biological risk factors for cervical cancer including restoring and maintaining healthy vaginal microbiota, pH, and mucosal function, thereby preventing disturbed immunity and inflammation caused by dysbiosis and mucosal microtrauma. The purpose of this study is to provide a quantitative perception evaluation of the acceptability of PreBioGyn and its applicator system.

The objectives of this study are to:

1. Perform a quantitative sensory evaluation to determine the topical acceptability of PreBioGyn, as well as receive qualitative feedback on the gel, as compared to competitive products.
2. Obtain quantitative and qualitative feedback regarding acceptability of the PreBioGyn applicator compared to those for existing competitive products.

These Study Objectives do not involve actual intravaginal use of the product. Rather, this activity will involve presentation of the products in a forearm and finger-touch sensory evaluation, and the answering of questions related to this perceptual evaluation.

Study Design:

This is a randomized, single-blind, cross-over study that will include 42 women.

Study Procedures and Methods:

Quantitative sensory evaluation and qualitative feedback to determine the acceptability of the prebiotic vaginal gel (PreBioGyn) as compared to competitive products

Summary:

Quantitative evaluation of PreBioGyn and two competitive vaginal pH buffer-gels will be performed. The four key qualitative parameters to be evaluated are slipperiness, tackiness, appearance, and smell. These parameters are key functional outcomes for the final PreBioGyn formula. Qualitative feedback and likelihood of use for each gel will also be collected and scored.

1. Quantitative Assessment of Slipperiness and Tackiness ("lubricity").

   Quantitative perceptual lubricity (slipperiness and tackiness) will be determined using a standardized methodology wherein participants discriminate differences between the PreBioGyn and two competitive products, versus positive and negative anchor products. Products are evaluated on the skin (forearm area) ex vivo.

   Participants will each receive the positive and negative anchors, then the three gel products, on three different 4-cm circular forearm sites. The order of the gels, and the circle to which it was applied, will be determined randomly based on a computer-generated randomization table. Each treatment is replicated twice. Participants will be blinded to the specific products used.

   Fingers and circles will be wiped with a low-residue baby-wipe and paper towel. The investigator dispenses 0.2 ml of the sample into the center of the circle previously drawn on the forearm. The sample is rubbed in a circle using the index finger at a rate of 2 revolutions per second for 15 seconds and followed with another 45 seconds (60 second time point). A metronome is set at 120 bpm and played to standardize the manipulation rate.

   At time points 15 and 60 seconds, slipperiness is evaluated using a visual analog scale (VAS). The two ends of the visual analog scale are anchored by the phrases "not slippery" and "very slippery." The participant is asked to make a mark on the VAS at the point of their slipperiness assessment between the two anchors. Prior to study gel measurements, participants will perform evaluations on two products representing the negative anchor "not slippery" (lanolin) and positive anchor "very slippery" (Gun Oil™ lubricant).

   At the 60-second time point, and after the slipperiness score is recorded, subjects will assess tackiness by tapping their finger up and down for 5 seconds on the skin in the circle just used to assess slipperiness.

   Tackiness is evaluated using the visual analog scale. The two ends of the visual analog scale are anchored by the phrases "Not tacky or sticky" and "very tacky or sticky." The focus group participant is asked to make a mark on the VAS at the point of their tackiness assessment between the two anchors. Prior to study gel measurements, participants will perform evaluations on two products representing the anchors of "very tacky" (lanolin) and "not tacky" (Gun Oil® lubricant). The degree of slipperiness and tackiness is determined by measuring the distance of the participants mark on the visual analog scale from the left baseline.
2. Qualitative Assessment of Appearance and Smell and Overall Perception.

   Study participants will be asked to rate the appearance and smell of the PreBioGyn and competitive products following the end of the quantitative assessment period. The traditional nine-point hedonic scale will be used to assess the degree of liking or disliking of each gel's smell and appearance. The reliability, validity and discriminative ability of the scale has been proven in food, cosmetic, and personal care product acceptance tests.

   Two milliliters (2 ml) of each lubricant will be dispensed from a prefilled syringe onto a small clear plastic petri dish. The order of the gel will be determined randomly based on a computer-generated randomization table. Each treatment is replicated twice. Participants will be blinded to the product identity. Subjects will be asked to observe the gels under good lighting, smell the gels from a distance of approximately 2-5 cm from the end of their nose, and then rate each gel on the Hedonic scale. Finally, open-ended feedback on the gels, including likelihood of use as a proposed product to decrease cervical cancer risk, will occur using the "I Like, I Wish, What If" method to gather participant contributions.
3. Quantitative and Qualitative Feedback Regarding Acceptability of the PreBioGyn Applicator Compared to Competitive Products.

Women will rank the PreBioGyn applicator versus that of competitive products in a 9-point Hedonic scale for acceptability of the applicator look and feel; the usability for preparing the applicator for dosing, and the usability to expel the gel (table-top). Finally, the overall reaction to the concept of inserting each applicator vaginally will be rated, as well as a 5-point Likert-scale rating of likelihood of future use of each product to reduce cervical cancer risk. Finally, open-ended feedback on the applicators will occur using the "I Like, I Wish, What If" method to gather participant contributions.

ELIGIBILITY:
Inclusion Criteria:

* Female
* hrHPV positive
* 30 years of age or older
* Have not received the HPV vaccine
* Not pregnant or nursing
* Medicaid eligible

Exclusion Criteria:

* history of skin irritation and/or allergic skin reactions

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Sensory perceptual characteristics of gels based on forearm testing | 1 hour
User acceptability of gel delivery system | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Ellington, PhD, Principal Investigator — Glyciome, LLC
Locations (2):
- Brigham and Women'S Hospital, Boston, Massachusetts, United States
- University of Puerto Rico Medical Sciences, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No